CLINICAL TRIAL: NCT02135796
Title: ICU Echocardiography in Resuscitation of Sepsis and Septic Shock
Brief Title: Echocardiography in Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1009957
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Septic Shock; Severe Sepsis
Keywords: Septic Shock; Severe Sepsis; ICU
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sepsis/Septic Shock: Individuals who are admitted to the Intensive Care Unit (ICU) with an infection called Sepsis or Septic Shock. This group will receive transthoracic echocardiography as part of the study.
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography

SUMMARY:
BACKGROUND: Echocardiography can provide evaluation of right or left ventricular dysfunction and volume status during resuscitation of patients with sepsis and septic shock and guide intravenous vasopressor and fluid therapy. While there are numerous echocardiographic studies regarding cardiac function and volume status in patients with established shock, there are none that describe these during the early resuscitation of septic shock.

The study objective is to correlate echocardiographic findings with clinical parameters and net fluid balance measured during the early resuscitation of critically ill patients with sepsis and septic shock.

Aim 1) correlate echocardiographic findings of cardiac function with physiologic markers in the early hours of resuscitation

Aim 2) correlate cardiac function and fluid status with clinical outcomes

Aim 3) evaluate the change in cardiac function over time in patients with sepsis and septic shock

Aim 4) evaluate long term clinical outcomes for patients with sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

- at least 13 years of age

SEPSIS PATIENTS:

Sepsis patients must have

1. Suspected or confirmed infection

   AND
2. Organ dysfunction as defined by a SOFA >= 2 above baseline (if no baseline data available, SOFA assumed to be 0)

OR

SEPTIC SHOCK PATIENTS:

AFTER INFUSION OF 20ML/KG CRYSTALLOID OR EQUIVALENT, Septic shock patients must have

1. Suspected or confirmed infection

   AND
2. Lactate > 2 mmol/L

   AND
3. Receiving vasopressors

   * Enrollment of patients should occur within 8 hours of meeting criteria for severe sepsis or septic shock if it is required that a research only TTE be performed in the 0-6 hours after ICU admission. If a clinical TTE is performed in this timeframe, patients may be enrolled up to 24 hours after ICU admission.

Exclusion Criteria:

None.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to an Intensive Care Unit (ICU) with an initial diagnosis of severe sepsis or septic shock.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2008-10; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Correlate echo findings and markers of resuscitation | Within 12 hours of Intensive Care Unit admission
  Correlate echocardiographic findings of cardiac function with physiologic markers in the early hours of resuscitation. Specifically, cardiac markers will be analyzed in relation to cardiac function, including ejection fraction, strain, and diastolic function, and correlate these with several clinical parameters, including receipt of fluid, vasopressors, mechanical ventilation, and septic cardiomyopathy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lanspa, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No